CLINICAL TRIAL: NCT02292706
Title: A Registry for Subjects With Cirrhosis Who Achieve a Sustained Virologic Response Following Treatment With a Sofosbuvir-Based Regimen Without Interferon for Chronic Hepatitis C Infection
Brief Title: A Registry for Participants With Cirrhosis Who Achieve a Sustained Virologic Response Following Treatment With a Sofosbuvir-Based Regimen Without Interferon for Chronic Hepatitis C Infection
Status: Terminated | Type: Observational
Why Stopped: The study stopped early because the study objectives were met.
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Other Study IDs: GS-US-337-1431; 2014-001249-26 (EudraCT Number)
Record Dates: First submitted 2014-11-13; First posted 2014-11-17 (Estimated); Results first posted 2023-10-04 (Actual); Last update posted 2023-10-04 (Actual); Status verified 2022-12

CONDITIONS: Hepatitis C Virus Infection
Keywords: HCV Cirrhosis registry; Cirrhosis; Hepatitis C
MeSH Terms: conditions — Hepatitis C; Fibrosis | interventions — Sofosbuvir; Ribavirin; ledipasvir, sofosbuvir drug combination; sofosbuvir-velpatasvir drug combination; sofosbuvir velpatasvir voxilaprevir drug combination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (8):
- SOF+RBV: Participants who were previously treated with sofosbuvir (SOF) along with ribavirin (RBV) will be followed up to 5 years.
  Interventions: Drug: Sofosbuvir; Drug: Ribavirin
- LDV/SOF: Participants who were previously treated with ledipasvir/sofosbuvir (LDV/SOF) will be followed up to 5 years.
  Interventions: Drug: LDV/SOF
- LDV/SOF+RBV: Participants who were previously treated with LDV/SOF along with ribavirin will be followed up to 5 years.
  Interventions: Drug: Ribavirin; Drug: LDV/SOF
- SOF/VEL: Participants who were previously treated with sofosbuvir/velpatasvir (SOF/VEL) will be followed up to 5 years.
  Interventions: Drug: SOF/VEL
- SOF/VEL+RBV: Participants who were previously treated with SOF/VEL along with RBV will be followed up to 5 years.
  Interventions: Drug: Ribavirin; Drug: SOF/VEL
- SOF/VEL/VOX: Participants who were previously treated with sofosbuvir/velpatasvir/voxilaprevir (SOF/VEL/VOX) with or without RBV will be followed up to 5 years.
  Interventions: Drug: Ribavirin; Drug: SOF/VEL/VOX
- Other SOF-Based: Participants who previously received other SOF based regimen will be followed up to 5 years.
  Interventions: Drug: Other SOF-Based Regimen
- Enrolled From Ineligible Parent Treatment Group: Participants were enrolled from ineligible parent treatment group.
  Interventions: Other: Ineligible parent treatment

INTERVENTIONS:
Drug: Sofosbuvir — Exposure of interest for participants who received sofosbuvir in a previous Gilead study for chronic HCV infection.
  Other Names: Sovaldi®; GS-7977; PSI-7977
  Groups: SOF+RBV
Drug: Ribavirin
  Groups: LDV/SOF+RBV; SOF+RBV; SOF/VEL+RBV; SOF/VEL/VOX
Drug: LDV/SOF — Exposure of interest for participants who received LDV/SOF in a previous Gilead study for chronic HCV infection.
  Other Names: Harvoni®
  Groups: LDV/SOF; LDV/SOF+RBV
Drug: SOF/VEL — Exposure of interest for participants who received SOF/VEL in a previous Gilead study for chronic HCV infection.
  Other Names: Epclusa®
  Groups: SOF/VEL; SOF/VEL+RBV
Drug: SOF/VEL/VOX — Exposure of interest for participants who received SOF/VEL/VOX in a previous Gilead study for chronic HCV infection.
  Other Names: Vosevi®
  Groups: SOF/VEL/VOX
Drug: Other SOF-Based Regimen — The other SOF-based regimens may have included the following:
  * BMS-790052 (Daclatasvir) + GS-7977 (SOF) with or without RBV
  * LDV/SOF + GS-9669, GS-7977 (SOF) + with or without RBV + TMC-435 (Simeprevir)
  * LDV/SOF + Vedroprevir (VDV), LDV/SOF + GS-9669 (250 mg and 500 mg)
  * LDV/SOF + VDV + RBV
  * Simeprevir + SOF
  * TMC-435 (Simeprevir) + VEL/SOF
  Groups: Other SOF-Based
Other: Ineligible parent treatment — Participants were enrolled from ineligible parent treatment group.
  Groups: Enrolled From Ineligible Parent Treatment Group

SUMMARY:
The primary objective of this registry study is to assess the durability of sustained virologic response (SVR) and clinical progression or regression of liver disease including the incidence of hepatocellular carcinoma following SVR in participants with cirrhosis after treatment with a sofosbuvir-based regimen for HCV infection.

ELIGIBILITY:
Key Inclusion Criteria:

* Willing and able to provide written informed consent
* Have either previously participated in a Gilead-sponsored HCV study and received a sofosbuvir-containing regimen without interferon OR at pre-selected sites only, have received an all-oral SOF-based regimen outside a clinical study. These individuals must have documentation of the regimen, start and end of treatment dates (month and year), and of having achieved SVR12.
* Have achieved SVR either in a Gilead-sponsored study, as defined in the treatment protocol OR for individuals who enroll after receiving an all-oral SOF-based regimen outside a clinical study, SVR will be defined as HCV RNA < lower limit of quantification (LLOQ) approximately 12 weeks following last dose of treatment.
* Have liver cirrhosis, as defined in the treatment protocol, and have not had a liver transplant after receiving a SOF-containing regimen OR individuals who enroll after receiving an all-oral SOF-based regimen outside a clinical study, will have had cirrhosis confirmed prior to initiation of HCV treatment.

Key Exclusion Criteria:

* Individuals planning to initiate a new course of HCV therapy, including approved products and any investigational agents, during the course of this Registry
* History of clinically-significant illness or any other major medical disorder that may interfere with the follow-up, assessments, or compliance with the protocol

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with cirrhosis who have achieved an SVR after receiving a SOF-based regimen without interferon (IFN) while participating in a Gilead-sponsored HCV study. In addition, participants with cirrhosis who have achieved SVR after an all-oral SOF-based regimen outside a clinical study may be eligible to enroll in this registry at sites preselected by Gilead.
Sampling Method: Non-Probability Sample
Enrollment: 1609 (Actual)
Dates: Start 2014-12-29 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (138):
- United States (77):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Scripps Clinic Medical Group, La Jolla, California
  - V.A. Long Beach Medical Center, Long Beach, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - Kaiser Permanente Medical Center, Los Angeles, California
  - Tarrant County ID Associates, Los Angeles, California
  - The Liver Center, Pasadena, California
  - Inland Empire Liver Foundation, Rialto, California
  - University of California, Davis Medical Center, Sacramento, California
  - Kaiser Permanente, San Diego, California
  - Medical Associates Research Group, San Diego, California
  - Quest Clinical Research, San Francisco, California
  - University of California at San Francisco Medical Center, San Francisco, California
  - Stanford University, Stanford, California
  - University of Colorado, Aurora, Colorado
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - Whitman-Walker Health, Washington D.C., District of Columbia
  - UF Hepatology Research at CTRB, Gainesville, Florida
  - Borland-Groover Clinic, Jacksonville, Florida
  - University of Miami Miller School of Medicine, Miami, Florida
  - Orlando Immunology Center, Orlando, Florida
  - Tampa General Hospital, Tampa, Florida
  - South Florida Center of Gastroenterology, Wellington, Florida
  - Atlanta Gastroenterology Associates, Atlanta, Georgia
  - Atlanta Medical Center, Atlanta, Georgia
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Gastrointestinal Specialists of Georgia, PC, Marietta, Georgia
  - Northwestern University, Chicago, Illinois
  - Indiana University, Indianapolis, Indiana
  - Indianapolis Gastroenterology Research Foundation, Indianapolis, Indiana
  - University of Kansas Medical Center Research Institute, Inc., Kansas City, Kansas
  - Delta Research Partners, Monroe, Louisiana
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Mercy Medical Center, Baltimore, Maryland
  - Digestive Disease Associates, PA, Catonsville, Maryland
  - Johns Hopkins Hospital/University, Lutherville, Maryland
  - Community Research Initiative of New England, Boston, Massachusetts
  - BIDMC Liver Center, Boston, Massachusetts
  - University of Michigan Medical Center, Ann Arbor, Michigan
  - Henry Ford Health System, Detroit, Michigan
  - University of Minnesota Medical Center, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Minnesota Gastroenterology, PA, Saint Paul, Minnesota
  - Kansas City Research Institute, LLC, Kansas City, Missouri
  - Saint Louis University, St Louis, Missouri
  - ID Care, Inc, Hillsborough, New Jersey
  - Southwest CARE Center, Santa Fe, New Mexico
  - Binghamton Gastroenterology Associates, PC, Binghamton, New York
  - North Shore Health Inc., Manhasset, New York
  - Columbia University Medical Center, New York, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - New York University Medical Center, New York, New York
  - Weill Cornell Medical College, New York, New York
  - Asheville Gastroenterology Associates, PA, Asheville, North Carolina
  - Carolinas Medical Center, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Cumberland Research Associates, LLC, Fayetteville, North Carolina
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - University of Pennsylvania Health System, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - University Gastroenterology, Providence, Rhode Island
  - Gastroenterology Center of the MidSouth, P.C., Germantown, Tennessee
  - Nashville Gastrointestinal Specialists, Inc., Nashville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - The North Texas Clinical Research Institute, Arlington, Texas
  - Baylor Endocrine Center, Dallas, Texas
  - North Texas Research Institute, Dallas, Texas
  - St. Luke's Episcopal Hospital, Houston, Texas
  - The Texas Liver Institute, San Antonio, Texas
  - Intermountain Medical Center, Murray, Utah
  - INOVA Fairfax Hospital, Annandale, Virginia
  - Bon Secours St. Mary's Hospital of Richmond, Newport News, Virginia
  - Digestive and Liver Disease Specialists, Norfolk, Virginia
  - Harborview Medical Center, Seattle, Washington
  - Virginia Mason Medical Center, Seattle, Washington
- Australia (11):
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - Kirby Institute, Sydney, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Royal Brisbane & Women's Hospital, Herston, Queensland
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - St Vincents Hospital Sydney, Fitzroy, Victoria
  - Austin Health, Heidelberg, Victoria
  - Monash Medical Centre Clayton Campus, Melbourne, Victoria
  - The Alfred Hospital, Prahran, Victoria
  - Fiona Stanley Hospital, Fremantle, Western Australia
  - Royal Perth Hospital, Perth, Western Australia
- Canada (7):
  - University of Calgary, Calgary, Alberta
  - GI Research Institute, Vancouver, British Columbia
  - Vancouver Infectious Disease Research and Care Centre, Vancouver, British Columbia
  - London Health Sciences Centre - University Campus, London, Ontario
  - University Health Network, Toronto, Ontario
  - CRCHUM, Montreal, Quebec
  - University of Alberta, Edmonton
- France (18):
  - Hôpital Pontchaillou, Rennes, Brittany Region
  - CHU Montpellier - Hopital St. Eloi, Montpellier, Languedoc-Rousillon
  - Hôpital Universitaire Dupuytren, Limoges, Limousin
  - Hopital Purpan, Toulouse, Midi-Pyrenees
  - Groupe Hospitalier Archet I Et II, Nice, Provence Alpes Cote D'Azu
  - Hopital Saint Joseph, Marseille, Provence-Alpes-Côte d'Azur Region
  - Hopital Haut Leveque, Bordeaux
  - CHU Estaing, Clermont-Ferrand
  - Hôpital Beaujon, Clichy
  - Hopital Henri Mondor, Créteil
  - CHU de Grenoble- Hopital Michallon, Grenoble
  - Hopital Cochin, Paris
  - Hopital Tenon, Paris
  - Hôpital de la Croix Rousse, Paris
  - Hôpitaux Universitaires de Strasbourg, Strasbourg
  - CHU de Nancy-Hopital Brabois Adulte, Vandœuvre-lès-Nancy
  - Hôpital Paul Brousse, Villejuif
  - Hopital de La Pitié-Salpêtrière, Paris, Île-de-France Region
- Germany (5):
  - Universitatsklinikum Koln, Cologne
  - Klinikum der Johann Wolfgang Goethe Universitat, Frankfurt am Main
  - Universitätsklinikum Hamburg-Eppendorf, Hamburg
  - Asklepios Klinik St. Georg, Hamburg
  - Technische Universität München, Mücheln
- Italy (4):
  - Azienda Ospedaliera Ospedale Niguarda Cà Granda, Milan
  - Fondazione IRCCS Cà Granda Ospedale Maggiore Policlinico, Milan
  - Ospedale Casa Sollievo Della Sofferenza IRCCS, San Giovanni Rotondo
  - Azienda Ospedaliera Città della Salute e della Scienza di Torino, Torino
- New Zealand (3):
  - Auckland Clinical Studies Ltd, Auckland, North Island
  - Waikato Hospital, Hamilton, North Island
  - Christchurch Hospital, Christchurch, South Island
- Fundacion de Investigation de Diego, San Juan, Puerto Rico
- Spain (5):
  - Hospital Universitario Puerta de Hierro Majadahonda, Majadahonda, Madrid
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Hospital Virgen de Valme, Seville
  - Hospital Universitari i Politecnic La Fe de Valencia, Valencia
- United Kingdom (7):
  - Barts Health NHS Trust, London, England
  - Kings College Hospital, London, England
  - St Georges University of London, London, England
  - North Manchester General Hospital, Manchester, England
  - Nottingham University Hospitals NHS Trust, Nottingham, England
  - Gartnavel General Hospital, Glasgow, Scotland
  - Queen Alexandra Hospital, Portsmouth

IPD SHARING:
Plan to Share IPD: Yes
Qualified external researchers may request IPD for this study after study completion. For more information, please visit our website at https://www.gileadclinicaltrials.com/transparency-policy/
Supporting Information: Study Protocol, SAP
Time Frame: 18 months after study completion
Access Criteria: A secured external environment with username, password, and RSA code.
URL: https://www.gileadclinicaltrials.com/transparency-policy/

REFERENCES:
- [Background] Dunn W, Koestler D, Ni L, Kersey K, Kreter B, Hammond K et al. Cirrhosis regression based on both Enhanced Liver Fibrosis (ELF) and Fibrotest after Direct-acting Hepatitis C therapeutics corresponds to a lower incidence rate of hepatocellular carcinoma below the cost-effective threshold for surveillance [Poster 1289]. The International Liver Congress™ EASL - European Association for the Study of the Liver (EASL); 2021 23-26 June.
- [Background] Fan R, Papatheodoridis G, Sun J, Innes H, Toyoda H, Xie Q, Mo S, Sypsa V, Guha IN, Kumada T, Niu J, Dalekos G, Yasuda S, Barnes E, Lian J, Suri V, Idilman R, Barclay ST, Dou X, Berg T, Hayes PC, Flaherty JF, Zhou Y, Zhang Z, Buti M, Hutchinson SJ, Guo Y, Calleja JL, Lin L, Zhao L, Chen Y, Janssen HLA, Zhu C, Shi L, Tang X, Gaggar A, Wei L, Jia J, Irving WL, Johnson PJ, Lampertico P, Hou J. aMAP risk score predicts hepatocellular carcinoma development in patients with chronic hepatitis. J Hepatol. 2020 Dec;73(6):1368-1378. doi: 10.1016/j.jhep.2020.07.025. Epub 2020 Jul 21. PMID 32707225
- [Background] Jacobson I, Muir AJ, Lawitz EJ, Gane E, Conway B, Ruane PJ, et al. Course of Cirrhosis Regression: Lessons From Patients With HCV Cirrhosis Following Successful Sofosbuvir-Based Treatment [Poster 537]. AASLD: The Liver Meeting® 2019, November 11-15.
- [Background] Mangia A, Lawitz E, Gane E Conway B, Ruane PJ, Abergel A, et al. Long-Term Follow-up of Patients with Chronic HCV Infection and Compensated or Decompensated Cirrhosis Following Treatment with Sofosbuvir-Based Regimens. The International Liver Congress™ EASL - European Association for the Study of the Liver (EASL); 2018 April 11-15.
- [Background] Muir AJ, Buti M, Nahass R, Agarwal K, Gane EJ, Strasser SI, et al. Long-term Follow-up of Patients With Chronic HCV Infection and Compensated or Decompensated Cirrhosis Following Treatment With Sofosbuvir-Based Regimens [Poster 880]. AASLD: The Liver Meeting® 2019, November 11-15.
- [Background] Reddy KR, Bourlière M, Agarwal K, Lawitz E, Osinusi A, Kersey K, et al. Sustained Viral Response Following Treatment With Direct-Acting Antiviral Agents for Chronic Hepatitis C and the Risk of Hepatocellular Carcinoma [Poster FRI-185]. The International Liver Congress™ EASL - European Association for the Study of the Liver (EASL); 2017 19-23 April.
- [Background] Reddy R, Muir A, Naggie S, Lawitz E, Gane E, Conway B et al. Noninvasive Tests of Fibrosis and Risk of Liver-Related Complications: Lessons From Patients With HCV Cirrhosis Following Successful Sofosbuvir-Based Treatment [Poster 452]. The International Liver Congress™ EASL - European Association for the Study of the Liver (EASL); 2020 27-29 August.
- [Background] Reddy R, Muir A, Naggie S, Lawitz E, Gane E, Conway B et al. Non-invasive tests of fibrosis and risk of liver-related complications: observations following successful sofosbuvir-based treatment in patients with HCV cirrhosis. J Hepatology 2020;73: S401-S652.
- [Derived] Younossi ZM, Racila A, Muir A, Bourliere M, Mangia A, Esteban R, Zeuzem S, Colombo M, Manns M, Papatheodoridis GV, Buti M, Chokkalingam A, Gaggar A, Nader F, Younossi I, Henry L, Stepanova M. Long-term Patient-Centered Outcomes in Cirrhotic Patients With Chronic Hepatitis C After Achieving Sustained Virologic Response. Clin Gastroenterol Hepatol. 2022 Feb;20(2):438-446. doi: 10.1016/j.cgh.2021.01.026. Epub 2021 Jan 22. PMID 33493697
- See also: Gilead Clinical Trials Website — https://www.gileadclinicaltrials.com/study/?id=GS-US-337-1431

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in Australia, Canada, France, Germany, Italy, New Zealand, Spain, the United Kingdom, and the United States.
Pre-assignment Details: 1609 participants were enrolled in the registry. 36 participants who were enrolled but did not meet the eligibility criteria (including 19 participants in the 'Enrolled from Ineligible Parent Treatment Group') were not included in the Full Analysis Set and Safety Analysis Set, and thus, are not included in the Baseline Characteristics, Outcome Measures and Serious and Other Adverse Event modules.
Groups:
- SOF+RBV: Participants who were previously treated with sofosbuvir (SOF) along with ribavirin (RBV) were followed up to 5 years.
- LDV/SOF: Participants who were previously treated with ledipasvir (LDV)/SOF were followed up to 5 years.
- LDV/SOF+RBV: Participants who were previously treated with LDV/SOF along with RBV were followed up to 5 years.
- SOF/VEL: Participants who were previously treated with SOF/velpatasvir (VEL) were followed up to 5 years.
- SOF/VEL+RBV: Participants who were previously treated with SOF/VEL along with RBV were followed up to 5 years.
- SOF/VEL/VOX: Participants who were previously treated with SOF/VEL/voxilaprevir (VOX) with or without RBV were followed up to 5 years.
- Other SOF-Based: Participants who previously received other SOF based regimen were followed up to 5 years.
Period: Overall Study
Arm/Group | SOF+RBV | LDV/SOF | LDV/SOF+RBV | SOF/VEL | SOF/VEL+RBV | SOF/VEL/VOX | Other SOF-Based | Enrolled From Ineligible Parent Treatment Group
Started | 95 | 277 | 265 | 374 | 100 | 338 | 141 | 19
Completed | 49 | 145 | 157 | 201 | 35 | 181 | 82 | 0
Not Completed | 46 | 132 | 108 | 173 | 65 | 157 | 59 | 19
Not completed — Lost to Follow-up | 20 | 44 | 24 | 61 | 21 | 52 | 25 | 0
Not completed — Withdrew consent | 15 | 56 | 43 | 36 | 13 | 51 | 20 | 0
Not completed — Death | 3 | 11 | 16 | 22 | 8 | 17 | 3 | 0
Not completed — Study terminated by sponsor | 0 | 9 | 4 | 21 | 11 | 13 | 3 | 0
Not completed — Investigator's discretion | 4 | 9 | 7 | 11 | 4 | 10 | 1 | 0
Not completed — Liver transplant | 1 | 1 | 11 | 16 | 5 | 6 | 5 | 0
Not completed — Enrolled but not met eligibility criteria | 1 | 2 | 2 | 2 | 2 | 6 | 2 | 19
Not completed — Subject terminated by sponsor | 1 | 0 | 0 | 2 | 1 | 0 | 0 | 0
Not completed — Missing | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0
Not completed — Virologic relapse or reinfection | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set included participants who met all inclusion criteria and did not meet any of the exclusion criteria, and with at least one post-enrollment visit measurement available.
Groups:
- SOF+RBV: Participants who were previously treated with SOF along with RBV were followed up to 5 years.
- LDV/SOF: Participants who were previously treated with SOF/LDV were followed up to 5 years.
- LDV/SOF+RBV: Participants who were previously treated with SOF/LDV along with RBV were followed up to 5 years.
- SOF/VEL: Participants who were previously treated with SOF/VEL were followed up to 5 years.
- SOF/VEL/VOX: Participants who were previously treated with SOF/VEL/VOX with or without RBV were followed up to 5 years.
- Total: Total of all reporting groups
Arm/Group | SOF+RBV | LDV/SOF | LDV/SOF+RBV | SOF/VEL | SOF/VEL+RBV | SOF/VEL/VOX | Other SOF-Based | Total
Number analyzed (Participants) | 94 | 275 | 263 | 372 | 98 | 332 | 139 | 1573
Age, Continuous [Mean (Standard Deviation); unit: years] | 56 (7.4) | 60 (7.8) | 60 (7.2) | 58 (7.3) | 58 (6.9) | 59 (7.6) | 59 (8.1) | 59 (7.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 94 | 83 | 115 | 28 | 87 | 55 | 497
  Male | 59 | 181 | 180 | 257 | 70 | 245 | 84 | 1076
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 87 | 239 | 219 | 331 | 90 | 281 | 117 | 1364
  Not Hispanic or Latino | 7 | 34 | 41 | 35 | 8 | 49 | 22 | 196
  Unknown or Not Reported | 0 | 2 | 3 | 6 | 0 | 2 | 0 | 13
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 82 | 230 | 234 | 324 | 86 | 292 | 117 | 1365
  Race: Black | 3 | 40 | 19 | 25 | 5 | 26 | 20 | 138
  Race: Asian | 7 | 3 | 4 | 17 | 5 | 8 | 0 | 44
  Race: American Indian or Alaska Native | 1 | 0 | 2 | 4 | 0 | 1 | 1 | 9
  Race: Unknown or Not Reported | 0 | 2 | 2 | 2 | 0 | 2 | 1 | 9
  Race: Native Hawaiian or Other Pacific Islander | 1 | 0 | 1 | 0 | 1 | 2 | 0 | 5
  Race: Other | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  New Zealand | 4 | 3 | 13 | 9 | 4 | 30 | 3 | 66
  Canada | 5 | 0 | 5 | 24 | 0 | 16 | 0 | 50
  United States | 50 | 221 | 166 | 241 | 76 | 228 | 136 | 1118
  Italy | 1 | 2 | 13 | 10 | 0 | 0 | 0 | 26
  United Kingdom | 14 | 0 | 4 | 22 | 0 | 9 | 0 | 49
  Australia | 14 | 0 | 12 | 24 | 2 | 13 | 0 | 65
  France | 0 | 46 | 32 | 20 | 0 | 24 | 0 | 122
  Germany | 1 | 3 | 3 | 7 | 0 | 12 | 0 | 26
  Spain | 5 | 0 | 15 | 15 | 16 | 0 | 0 | 51

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Maintaining Sustained Virologic Response (SVR) at Week 240
Description: SVR at Week 240 was defined as HCV RNA< lower limit of quantification (LLOQ i.e., 15 or 25 international units per milliliter [IU/mL]) or last available HCV RNA< LLOQ with no subsequent follow-up values at Week 240 after enrollment in this registry study. Percentage of participants who maintained SVR status by Week 240 was estimated using a Kaplan-Meier model.
Time Frame: Week 240
Population: Full Analysis Set included all participants who met all inclusion criteria and did not meet any of the exclusion criteria, and with at least one post-enrollment visit measurement available.
Measure: Number; unit: percentage of participants
Groups:
- LDV/SOF: Participants who were previously treated with LDV/SOF were followed up to 5 years.
Arm/Group | SOF+RBV | LDV/SOF | LDV/SOF+RBV | SOF/VEL | SOF/VEL+RBV | SOF/VEL/VOX | Other SOF-Based
Number analyzed (Participants) | 94 | 275 | 263 | 372 | 98 | 332 | 139
percentage of participants | 98.9 | 100 | 99.6 | 99.7 | 100 | 99.6 | 100

2. Primary Outcome: Percentage of Participants With Any Liver-Associated Events
Description: The percentage of participants with any liver-associated events since registry start (enrollment) through Week 240 was estimated using a Kaplan-Meier model.
Time Frame: Enrollment up to 240 weeks
Population: Participants in Full Analysis Set who did not develop liver-associated event prior to entering the registry were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | SOF+RBV | LDV/SOF | LDV/SOF+RBV | SOF/VEL | SOF/VEL+RBV | SOF/VEL/VOX | Other SOF-Based
Number analyzed (Participants) | 89 | 259 | 254 | 350 | 81 | 326 | 133
percentage of participants | 18.7 | 15.0 | 24.8 | 18.1 | 37.6 | 16.1 | 18.2

3. Primary Outcome: Percentage of Participants Who Developed Hepatocellular Carcinoma (HCC) Through Week 240
Description: Participants with de novo HCC since registry start were defined as participants who had not been identified with HCC prior to registry start and only had HCC since registry start. The percentage of participants who developed de novo HCC through Week 240 was estimated using a Kaplan-Meier model.
Time Frame: Enrollment up to 240 weeks
Population: Participants in the Full Analysis Set with no HCC prior to this registry study were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | SOF+RBV | LDV/SOF | LDV/SOF+RBV | SOF/VEL | SOF/VEL+RBV | SOF/VEL/VOX | Other SOF-Based
Number analyzed (Participants) | 92 | 273 | 259 | 367 | 98 | 330 | 138
percentage of participants | 11.8 | 5.01 | 10.8 | 10.8 | 15.3 | 12.4 | 11.2

4. Secondary Outcome: Number of Participants With Detectable HCV RNA Due to Re-emergence of Pre-existing Virus Through Week 240
Time Frame: Enrollment up to 240 weeks
Population: Participants in Full Analysis Set were analyzed.
Measure: Count of Participants; unit: Participants
Groups:
- LDV/SOF+RBV: Participants who were previously treated with either LDV/SOF along with RBV were followed up to 5 years.
Arm/Group | SOF+RBV | LDV/SOF | LDV/SOF+RBV | SOF/VEL | SOF/VEL+RBV | SOF/VEL/VOX | Other SOF-Based
Number analyzed (Participants) | 94 | 275 | 263 | 372 | 98 | 332 | 139
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0

5. Secondary Outcome: Number of Participants With Detectable HCV Resistance Mutations Through Week 240
Time Frame: Enrollment up to 240 weeks
Population: Participants in Full Analysis Set were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | SOF+RBV | LDV/SOF | LDV/SOF+RBV | SOF/VEL | SOF/VEL+RBV | SOF/VEL/VOX | Other SOF-Based
Number analyzed (Participants) | 94 | 275 | 263 | 372 | 98 | 332 | 139
Participants | 0 | 0 | 1 | 0 | 0 | 1 | 0

6. Secondary Outcome: Number of Participants With Detectable HCV RNA Due to Re-infection Through Week 240
Description: Reinfection was defined as HCV RNA > LLOQ on 2 samples collected at least 1 week apart with a different virus than that present prior to treatment baseline in the parent study.
Time Frame: Enrollment up to 240 weeks
Population: Participants in Full Analysis Set were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | SOF+RBV | LDV/SOF | LDV/SOF+RBV | SOF/VEL | SOF/VEL+RBV | SOF/VEL/VOX | Other SOF-Based
Number analyzed (Participants) | 94 | 275 | 263 | 372 | 98 | 332 | 139
Participants | 0 | 0 | 0 | 1 | 0 | 1 | 0

ADVERSE EVENTS:
Time Frame: All-Cause Mortality and Adverse Events (AEs): From enrollment up to maximum duration of 5 years
Description: All-Cause Mortality: Included participants who signed informed consent and enrolled into study.
  AEs: Included all participants who met all inclusion criteria and did not meet any of exclusion criteria, and with at least one post-enrollment visit measurement available; no participants were included in 'Enrolled from Ineligible Parent Treatment Group'. No study treatments were given to study participants; thus, reported adverse events refer to AEs related to study procedures.
Arm/Group | SOF+RBV | LDV/SOF | LDV/SOF+RBV | SOF/VEL | SOF/VEL+RBV | SOF/VEL/VOX | Other SOF-Based | Enrolled From Ineligible Parent Treatment Group
All-Cause Mortality (participants affected / at risk) | 3/95 | 11/277 | 16/265 | 22/374 | 8/100 | 17/338 | 3/141 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/94 | 0/275 | 0/263 | 0/372 | 0/98 | 0/332 | 0/139 | 0/0
Other Adverse Events (participants affected / at risk) | 0/94 | 4/275 | 1/263 | 1/372 | 0/98 | 1/332 | 1/139 | 0/0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SOF+RBV (N=94) | LDV/SOF (N=275) | LDV/SOF+RBV (N=263) | SOF/VEL (N=372) | SOF/VEL+RBV (N=98) | SOF/VEL/VOX (N=332) | Other SOF-Based (N=139) | Enrolled From Ineligible Parent Treatment Group (N=0)
Vessel puncture site haematoma (General disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0
Incision site rash (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Post procedural complication (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Procedural complication (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Procedural dizziness (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years

DOCUMENTS (2):
  • Study Protocol (2017-06-01): https://cdn.clinicaltrials.gov/large-docs/06/NCT02292706/Prot_000.pdf
  • Statistical Analysis Plan (2022-04-13): https://cdn.clinicaltrials.gov/large-docs/06/NCT02292706/SAP_001.pdf